CLINICAL TRIAL: NCT00848822
Title: Sleep and Glucose Regulation in Youth With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Priti Patel, M.D., University of Arizona
Other Study IDs: 08-1108-01
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Type 1 Diabetes Mellitus; Sleep
Keywords: Pediatrics; Sleep; Glucose regulation; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to look at how sleep affects glucose values in children with Type 1 Diabetes Mellitus. It will also evaluate if glucose is affected by times of day due to the body's own internal rhythm also known as the circadian rhythm.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is one of the most prevalent chronic pediatric diseases, affecting 2.80 cases per 1000 youth between the ages of 10 and 19. Since the crux of diabetes management is glucose regulation, any further challenges such as stress and/or poor sleep may make glucose regulation even more difficult. Mounting evidence supports the association between inadequate sleep and obesity as well as metabolic syndrome. Despite emerging findings supporting that total sleep time (TST) may contribute to the risk of obesity and/or metabolic complications, less research has been focused on Type 1 Diabetes Mellitus (T1DM) and on other sleep parameters.

Participants will have a Continuous Glucose Monitor (CGM) and actigraph placed which they will wear for 5 days. At the end of the 5 days, they will return the glucose meter, CGM, and actigraph to a clinic staff or research team member to download their data. They will provide us with a glucose log that contains the glucose levels obtained from a fingerstick capillary glucose meter. In this log, participants will also record their activities, meals, and insulin administered. They will also provide us with a sleep diary. In addition, participants will have the option for the child to undergo polysomnography (sleep study) for one night in their home or two nights in the sleep lab.

ELIGIBILITY:
Inclusion Criteria:

* Type I Diabetes Mellitus
* Age of 10-16 year old

Exclusion Criteria:

* Significant Developmental Delay
* Any other condition that in the opinion of the medical treatment team would interfere with his/her ability to participate

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pariticipants will be recruited from the Angel Clinic for Children with Diabetes and Endocrine Disorders which is part of University Medical Center in Tucson, Arizona
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
This study could help find if there are particular times of day or times during sleep that change glucose the most. | 12 months

SECONDARY OUTCOMES:
This study may help make recommendations about the best time to test glucose values and better help children with Type 1 Diabetes Mellitus control their glucose levels. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Priti G Patel, M.D., Principal Investigator — University of Arizona; Michelle Perfect, PhD, Principal Investigator — Univeristy of Arizona
Locations (1):
- Steele Research Memorial Foundation, Angel Clinic for Children with Diabetes and Endocrine Disorders, Tucson, Arizona, United States

REFERENCES:
- [Background] SEARCH for Diabetes in Youth Study Group; Liese AD, D'Agostino RB Jr, Hamman RF, Kilgo PD, Lawrence JM, Liu LL, Loots B, Linder B, Marcovina S, Rodriguez B, Standiford D, Williams DE. The burden of diabetes mellitus among US youth: prevalence estimates from the SEARCH for Diabetes in Youth Study. Pediatrics. 2006 Oct;118(4):1510-8. doi: 10.1542/peds.2006-0690. PMID 17015542
- [Background] Matyka KA, Crawford C, Wiggs L, Dunger DB, Stores G. Alterations in sleep physiology in young children with insulin-dependent diabetes mellitus: relationship to nocturnal hypoglycemia. J Pediatr. 2000 Aug;137(2):233-8. doi: 10.1067/mpd.2000.107186. PMID 10931417
- [Background] Pillar G, Schuscheim G, Weiss R, Malhotra A, McCowen KC, Shlitner A, Peled N, Shehadeh N. Interactions between hypoglycemia and sleep architecture in children with type 1 diabetes mellitus. J Pediatr. 2003 Feb;142(2):163-8. doi: 10.1067/mpd.2003.66. PMID 12584538
- [Background] Taras H, Potts-Datema W. Sleep and student performance at school. J Sch Health. 2005 Sep;75(7):248-54. doi: 10.1111/j.1746-1561.2005.00033.x. PMID 16102087